CLINICAL TRIAL: NCT02313038
Title: Prospective Assessment of Efficacy and Safety of Drug Eluting Stents
Acronym: PEACE-DES
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: MOST-2013BAI17B00
Record Dates: First submitted 2014-02-05; First posted 2014-12-09 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; Percutaneous Coronary Intervention; Drug Eluting Stents
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — A venous blood sample of 20mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage for future genetic studies; A urine samples of 40mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary heart disease (CHD) pose a serious health threat to population. PCI using drug eluting stents (DES), as a well-proved and booming measure in CHD management, is invasive and of high cost, however the knowledge about the real-life DES use and the efficacy and safety in China is limited. By consecutively recruiting first-ever PCI patients in 30 geographically representative highest-rank hospitals, this study will examine the prognosis in groups with different brands of DES, and various real-life factors, that may affect patients recovery after the procedure. Evidence for clinical practice and health resource allocation will be established based on the findings, to improve patients outcomes in future finally.

DETAILED DESCRIPTION:
In this study, 6000 patients who underwent the first-ever drug eluting stents (DES) deployment during the index hospitalization will be consecutively recruited in 30 tertiary hospitals scattered all over China. At study entry, participants will be interviewed during their index hospitalization, to collect information about symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. And CAG imaging will be reviewed by national and international expert panels. At 1 month, 6 month, and 12 month after discharge, participants will return to the clinic for follow up visits, a face-to-face interview will be conducted to get information about clinical events, symptoms, functioning, quality of life, and medical care during the recovery period. At 1-Month and 12-Month follow-up visit, blood and urine sample will be collected. Participants' blood samples will be stored for future biologic and genetic studies. This study will examine the prognosis in groups with different brands of DES, and various real-life factors, that may affect patients recovery after the procedure. Evidence for clinical practice and health resource allocation will be established based on the findings, to improve patients outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* At least one DES is implanted successfully in the procedure
* Only one of the five major brands of DES is used in the procedure

Exclusion Criteria:

* Prior stent implantation history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent the first-ever DES deployment during the index hospitalization were consecutively recruited.
Sampling Method: Non-Probability Sample
Enrollment: 6023 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Composite of major adverse cardiac events (MACE) | 1 year
  Composite of major adverse cardiac events (MACE) including death, myocardial infarction, and/or revascularization.

SECONDARY OUTCOMES:
Safety endpoint | 1 year
  Safety endpoint: stent thrombosis
Efficacy composite endpoints | 1 year
  Efficacy composite endpoints, including cardiac death, myocardial infarction (not clearly attributable to a nontarget vessel), and/or target lesion revascularization
Status of general health | 1 year
  Status of general health (SF-12)
Quality of life | 1 year
  Quality of life (EQ-5D)
Symptoms status | 1 year
  Symptoms status (SAQ)
Cost-effectiveness | 1 year
  Cost-effectiveness ratio: marginal cost (direct and indirect) per QALY increase, with homebred DES as the reference group

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, MD, PhD, Principal Investigator — China National Center for Cardiovascular Diseases; Harlan M Krumholz, MD, SM, Principal Investigator — Yale University
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China